CLINICAL TRIAL: NCT00046579
Title: Psychosocial Determinants of Nutrient Intake in Girls
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1184; R01HL071122 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To better understand the determinants of nutrient intake in black and white adolescent girls and to examine the effects of nutrient intake and eating behaviors on obesity, a significant risk factor for CVD.

DETAILED DESCRIPTION:
BACKGROUND:

Studies have documented the importance of eating behavior as a modifiable risk factor for the development of obesity and cardiovascular disease (CVD). The burden of obesity and CVD is not equally distributed in the population; women from ethnic minority populations are particularly likely to be obese and to have higher rates of CVD and stroke than white women.

DESIGN NARRATIVE:

The study determines the extent to which psychological and familial factors contribute to nutrient intake in black and white girls, beyond the well-established effects of ethnicity and socioeconomic factors. Specifically, the aims of the project are the following: 1) to provide a detailed developmental description of eating behaviors and nutrient intake in black and white girls and to examine the "clustering" of certain eating behaviors (e.g., skipping meals and snacking) into eating patterns; 2) to determine the clinical significance of eating behaviors and eating patterns by examining their contribution to nutrient intake and the development of obesity; 3) to examine the role of psychological and familial factors as determinants of eating behaviors, eating patterns, nutrient intake, and obesity in black and white girls. Capitalizing upon the availability of extensive data collected prospectively among an exceptionally well-maintained cohort of 2,379 black and white females over a 12-year period (from ages 9-10 to ages 21-23), the study applies innovative analytic procedures to further the scientific understanding of the determinants of nutrient intake and eating behaviors in adolescent girls. Participants were assessed annually for ten years as part of the National Heart, Lung and Blood Institute Growth and Health Study (NGHS) with measurements of anthropometry, food intake, eating and weight related attitudes and behaviors and family cohesion. Parents also provided information about weight, eating, and family environment at two assessments. In a subsequent study with the same sample, structured clinical interviews were conducted to determine history of psychiatric disorders and risk factors for eating disorders. Adult weight was also measured.

ELIGIBILITY:
No eligibility criteria

Ages: 9 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2002-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Striegel-Moore — Wesleyan University